CLINICAL TRIAL: NCT03406754
Title: Multi-disciplinary Rehabilitation Program for Advanced Parkinson's Patients in the Community
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-17-TG-0745-CTIL
Record Dates: First submitted 2018-01-07; First posted 2018-01-23 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ezera LaMarpeh rehabilitation programs: Participation in a rehabilitation program for 8 weeks
  Interventions: Behavioral: rehabilitation programs

INTERVENTIONS:
Behavioral: rehabilitation programs — an 8-week multidisciplinary inpatient rehabilitation program

SUMMARY:
The present study examines the effectiveness of the rehabilitation program in the framework of the "Ezra LeMarpeh" project for Parkinson's patients. The Ezra LeMarpeh Association, founded by Rabbi A. E. Firer, provides assistance to the sick and needy. The site features a wide range of advanced, high quality rehabilitation devices, a unique hydrotherapy pool and associated accessories that enable the staff to provide the finest quality and most professional treatment. Before entering a rehabilitative program, each participant will arrive independently at the Ezra LeMarpeh Center for evaluation tests and will undergo comprehensive evaluation tests by the center's physiotherapist, including walking tests, balance tests, filling out questionnaires to assess Quality of life and disease severity. At the end of the program, the participants will be asked to repeat evaluation tests.

DETAILED DESCRIPTION:
Before entering a rehabilitation program, each participant will arrive independently at the "Ezra LeMarpeh" Center, at 24 Chida St., Bnei Brak. After a detailed explanation of the nature of the study, the participants will sign an informed consent form. The center's physiotherapists will test walking abilities, motor functioning and abilities in activities of daily living (ADL).

Walking tests can include walking at a comfortable pace, walking while counting (dual tasking), walking at different speeds and more. The balance tests include standing on a small base, standing on one leg, standing with eyes closed, and more. During the tests participants will wear small, non-invasive sensors at the wrists, ankles, and lower back. These sensors include an accelerometers and a gyroscopes that can be used to quantify gait measures, such as gait velocity, step length and variability. Lower back sensors will be worn continuously for up to a week for everyday activity.

At the end of the program, the participants will be asked to repeat evaluation tests.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's disease, as defined in the UK Brain Bank criteria
2. Hoehn and Yahr stage I-III
3. Patients who are taking anti-Parkinson's drugs.
4. Participants who are in a stable medication regimen during the month preceding the study and are expected to remain in a permanent regime for the next 3 months.
5. Mini Mental State Exam (MMSE) score> 24
6. Able to walk independently for at least 5 minutes with or without support.

Exclusion Criteria:

1. Any neurological condition other than PD or orthopedic disease (eg after a stroke with neurological signs, MSA, Parkinsonism, PSP, etc.) that may impair normal walking and balance.
2. Significant cognitive impairment MMSE score<24
3. Any medical, surgical, and / or psychiatric condition which, in the opinion of the investigator, prevents the patient from completing all aspects of the research.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with parkinson's disease participated in rehabilitation program
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Immediate change in gait speed | Immediate at the end of the program (8 weeks)
  Gait speed will be assessed under usual and dual task conditions and while negotiating physical obstacles, using a sensorized 7 meter carpet (PKMAS) and wearable body fixed sensors. These measures will be compared to baseline performance.
Community ambulation | Immediate at the end of the program (8 weeks)
  Will be assessed using a body-worn small lightweight device (AX3 - continuous logging accelerometer) that will be worn by the subjects for 7 days to monitor ADL.

SECONDARY OUTCOMES:
Improve in motor function | Immediate at the end of the program (8 weeks)
  Timed Up & Go scores
Motor function | Immediate at the end of the program (8 weeks)
  UPDRS III scores

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Gurevich, MD, Principal Investigator — TASMC
Locations (2):
- Israel (2):
  - Laboratory for Gait and Neurodynamics, Tel Aviv Sourasky Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No